CLINICAL TRIAL: NCT00390156
Title: A Phase I Trial of Imatinib, Bevacizumab, & Metronomic Cyclophosphamide as Antiangiogenic Therapy in Refractory Metastatic Solid Tumors
Brief Title: Imatinib, Bevacizumab, and Cyclophosphamide in Patients With Refractory Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06991; 06991 (Other: UCSF); H9672-28868 (Other: UCSF CHR); CSTI571BUS245 (Other: Novartis)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Unspecified Adult Solid Tumor
Keywords: refractory; prior treatment; solid tumors; phase I; phase 1
MeSH Terms: interventions — Bevacizumab; Cyclophosphamide; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bevacizumab — 5 mg/kg
  Other Names: Avastin
Drug: cyclophosphamide — Current dose 50 mg
  Other Names: Cytoxan
Drug: imatinib — Current dose 400 mg
  Other Names: Gleevec

SUMMARY:
RATIONALE: Imatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bevacizumab and cyclophosphamide may also stop the growth of tumor cells by blocking blood flow to the tumor. Imatinib and bevacizumab may help cyclophosphamide work better by making tumor cells more sensitive to the drug. Giving cyclophosphamide once a day together with imatinib and bevacizumab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib when given together with bevacizumab and cyclophosphamide in treating patients with refractory metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of imatinib when given together with bevacizumab and metronomic cyclophosphamide in patients with refractory metastatic solid tumors.
* Determine the safety profile of this regimen in these patients.

Secondary

* Determine the effects of cyclophosphamide and bevacizumab on imatinib pharmacokinetics.
* Determine if patients treated with this regimen achieve plasma levels of cyclophosphamide that are predicted to be antiangiogenic.
* Determine the effects of this regimen on the number of circulating endothelial cells, endothelial progenitor cells, activated endothelial cells, and circulating tumor cells.
* Determine the effects of this regimen on parameters measured by CT scan perfusion (e.g., regional blood flow, blood volume, permeability-surface area product, and mean transit time).

OUTLINE: This is a nonrandomized, open-label, pilot, dose-escalation study of imatinib.

Patients receive oral cyclophosphamide and oral imatinib once daily on days 1-28 and bevacizumab IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor

  * Advanced or metastatic disease* NOTE: *With the exception of colorectal and lung cancer patients, all patients must receive approval from the insurance carrier that allows for coverage/payment of the study drug bevacizumab
* Refractory to standard therapy OR no standard therapy exists
* No advanced ovarian cancer or peritoneal carcinomatosis
* No metastases from any cancer causing significant ascites
* No lung malignancy with any of the following characteristics:

  * In close proximity to a major vessel
  * Centrally located
  * Cavitary
  * Squamous histology
  * Hemoptysis > ½ teaspoon per day

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Bilirubin < 2 mg/dL
* AST or ALT < 3 times upper limit of normal
* Creatinine < 2 mg/dL
* Urine protein:creatinine ratio ≤ 1.0
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to tolerate oral therapy
* No bleeding diatheses or coagulopathy
* No impairment of gastrointestinal (GI) function or GI disease that may affect or alter absorption of imatinib mesylate and/or cyclophosphamide (e.g., malabsorption syndrome, history of total gastrectomy/significant small bowel resection)
* No abdominal fistula, GI perforation, or intra-abdominal abscess within the past 6 months
* No uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg)
* No uncontrolled cardiovascular disease, including any of the following:

  * Coronary artery disease
  * Uncontrolled cardiac arrhythmia
  * Symptomatic congestive heart failure (i.e., New York Heart Association class II-IV)
  * Unstable angina pectoris
  * Clinically significant peripheral vascular disease
* No arterial thromboses within the past year, including any of the following:

  * Transient ischemic attack
  * Myocardial infarction
  * Cerebrovascular event
  * Unstable angina
  * Angina requiring medical or surgical intervention
  * Clinically significant peripheral artery disease
  * Any other arterial thromboembolic event
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No serious nonhealing wound, ulcer, or bone fracture
* No other active second malignancy except nonmelanoma skin cancer or cervical carcinoma in situ unless therapy has been completed and < 30% risk for relapse exists
* No active infection or known HIV infection
* No history of allergic reactions (≥ grade 3 or 4) to compounds of similar chemical or biologic composition to cyclophosphamide (i.e., alkylating agents)
* No history of noncompliance with medical regimens
* No known intolerance or hypersensitivity reaction to bevacizumab, imatinib mesylate, or cyclophosphamide
* No other significant medical illness, psychiatric illness, or social situation that, in the opinion of the investigator, would limit compliance with study requirements
* No inability to grant reliable informed consent

PRIOR CONCURRENT THERAPY:

* No major surgical procedure within the past 28 days or anticipated major surgery during study treatment except for placement of a venous access device or surgery for a diagnostic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of imatinib when given together with bevacizumab and metronomic cyclophosphamide | Safety data will be assessed after 3 patients and 6 patients complete 42 days of study treatment to determine whether to dose escalate to the next cohort.

SECONDARY OUTCOMES:
Pharmacokinetics of imatinib | After the last patient completes PKs on Cycle 1 Day 16
Safety of imatinib in combination with cyclophosphamide and bevacizumab | After all patients have completed study therapy. Safety data will be monitored throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Bergsland, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States